CLINICAL TRIAL: NCT04895761
Title: Phase Ib Study of Neoadjuvant DPX-Survivac, Aromatase Inhibition, and With/Without Radiotherapy or Cyclophosphamide in HR+HER2- Breast Cancer
Brief Title: Neoadjuvant DPX-Survivac Aromatase Inhibition, Radiotherapy or Cyclophosphamide in HR+HER2- Breast Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Providence Health & Services (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P2100-SUR-S11
Record Dates: First submitted 2021-05-17; First posted 2021-05-20 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Breast Cancer
Keywords: HR+/HER2
MeSH Terms: conditions — Breast Neoplasms | interventions — Letrozole; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Arm A: DPX-Survivac, Letrozole (Experimental): Letrozole 2.5 mg po daily, DPX-Survivac 0.25 mL SC week 2 and Week 5
  Interventions: Biological: DPX-Survivac; Drug: Letrozole 2.5mg
- Arm B: DPX-Survivac, Letrozole, Radiation (Experimental): Letrozole 2.5 mg po daily, XRT 10 Gy x 2, DPX-Survivac 0.25 mL SC week 2 and Week 5
  Interventions: Biological: DPX-Survivac; Drug: Letrozole 2.5mg; Radiation: XRT 10Gy x2
- Arm C: DPX-Survivac, Letrozole, cyclophosphamide (Experimental): Letrozole 2.5 mg po daily, cyclophosphamide 50 mg po BID, DPX-Survivac 0.25 mL SC week 2 and Week 5
  Interventions: Biological: DPX-Survivac; Drug: Letrozole 2.5mg; Drug: Cyclophosphamide 50mg

INTERVENTIONS:
Biological: DPX-Survivac — DPX is a novel formulation that when combined with target antigens acts to activate T cells. It is a lipid-based formulation that creates a long lasting depot at the site of injection, forcing an "active uptake" by antigen presenting cells (APCs). APCs traffic to regional lymph nodes where naïve T cells are activated, inducing strong and sustained immune responses. All arms will receive DPX-Survivac on weeks 2 and 5.
Drug: Letrozole 2.5mg — Aromatase inhibitor all arms will receive
  Other Names: Femara
Drug: Cyclophosphamide 50mg — oral chemotherapy used in the neoadjuvant setting for Arm C only
  Other Names: cytoxan
  Arms: Arm C: DPX-Survivac, Letrozole, cyclophosphamide
Radiation: XRT 10Gy x2 — Directed radiation at week 4 for Arm B only
  Arms: Arm B: DPX-Survivac, Letrozole, Radiation

SUMMARY:
The study seeks to establish the safety of neoadjuvant aromatase inhibitor with: DPX-Survivac, DPX-Survivac plus radiation, or DPX-Survivac with cyclophosphamide in stage I to III HR+HER2- breast cancer. There will be sequential enrollment into 3 arms with an anticipated N=6 participants per arm for N=18 participants in total. All participants will receive letrozole 2.5 mg daily during the 6 weeks of neoadjuvant therapy. Neoadjuvant therapy occurs weeks 1-6, with standard of care surgery taking place week 7 to 9.

DETAILED DESCRIPTION:
Women with hormone receptor positive, HER2-negative (HR+/HER2-) breast cancer with large tumors or positive lymph nodes have low response rates with neoadjuvant chemotherapy. Survivin is overexpressed in HR+HER2- breast cancer. Increasing tumor-specific Th1 immunity by administration of DPX-Survivac may alter the immune environment of these tumors. Radiation is a standard component of breast cancer therapy causing a reduction in local recurrences and improved breast cancer specific survival. Low dose cyclophosphamide can deplete regulatory T-cells without altering levels of effector T-cells. The investigators predict that combining a vaccine targeting Survivin, overexpressed in HR+HER2- tumors, with other immune modulating therapies such as radiation or low dose cyclophosphamide can enhance the efficacy of DPX-Survivac.

Primary Objective

1) Safety of neoadjuvant aromatase inhibitor with: DPX-Survivac, DPX-Survivac plus radiation, or DPX-Survivac with cyclophosphamide in stage I to III HR+HER2- breast cancer Secondary Objectives

1. Immunogenicity of each arm, assessed by IFN-γ ELISPOT in PBMC.
2. Immunogenicity of each arm, assessed by GEO-Mx digital spatial profiler evaluation of FFPE tissue and TCRβ evaluation for surviving-specific T cells in the tumor.

Exploratory Objectives

1. Evaluation of the % TIL in the biopsy specimen and at the time of surgery within/between arms
2. Evaluation of the Ki67 changes between the biopsy and at time of surgery within/between arms
3. Comparison of immunogenicity, TIL change, and Ki67 change across arms
4. Epitope spreading within/between arms
5. Evaluation of Triseq (germline, whole exome sequencing, and RNAseq) of the tumor immune environment within/between arms
6. Evaluation of immune environment using multi-parameter immunohistochemistry within/between arms
7. Evaluation by experimental MRI in arm that adds radiation
8. Evaluation of survivin-specific MHC-tetramer staining in PBMC

ELIGIBILITY:
Inclusion Criteria:

1. Patients must provide informed consent prior to any study-specific procedures and be able to understand and be willing to sign an informed consent document. Results of standard-of-care tests or examinations performed prior to obtaining informed consent and prior to treatment may be used for screening assessments rather than repeating such evaluations if within 30 day of day 1.
2. Women with resectable, non-metastatic breast cancer that is >1 cm, hormone receptor positive, HER2 negative, Ki67>10%.
3. HER2 negative is defined as:

   0-1+ HER2 expression by immunohistochemistry (IHC) OR Fluorescence in situ hybridization (FISH) negative OR HER2 2+ and FISH negative
4. Patients must be at least 28 days post systemic steroids prior to enrollment.
5. Patients must be at least 18 years of age.
6. Patients must have Eastern Cooperative Oncology Group (ECOG) Performance Status Score of ≤ 1
7. Adequate laboratory values within 30 days of enrollment defined as follows:

   1. White blood cell (WBC) ≥ 3000/mm3
   2. Hemoglobin (Hgb) ≥ 9 g/dL
   3. Neutrophil count ≥ 1500/mm3
   4. Lymphocyte count ≥ 1000/mm3
   5. Platelet count ≥ 75,000/mm3
   6. Serum creatinine ≤ 2.0 mg/dL or creatinine clearance > 60 ml/min
   7. Total bilirubin ≤ 1.5 mg/dL
   8. Aspartate aminotransferase (AST)/Serum glutamic oxaloacetic transaminase (SGOT) ≤ 2 times the ULN-
8. Patients must have recovered from major infections and, in the opinion of the investigator, do not have any significant active concurrent medical illnesses precluding protocol treatment.
9. The effects of DPX-Survivac on the developing human fetus are unknown. Women on the trial should be post-menopausal based on the NCCN definition of menopause
10. For patients in Arm B only, they must be able to undergo MR imaging as determined by treating physician using the standard Radiation Oncology MR screening process

Exclusion Criteria:

1. Patients may not be receiving any other investigational agents or on concurrent clinical trials while on during the clinical trial period.
2. History of allergic reactions attributed to compounds of similar chemical or biologic composition to DPX-Survivac.
3. Pregnant and pre-menopausal women are excluded from this study because to keep anti-endocrine therapy consistent between patients.
4. Known history of human immunodeficiency virus (HIV) infection, hepatitis B, or hepatitis C.
5. Uncontrolled autoimmune disease. Autoimmune disease allowed if controlled (with or without treatment) for the last 12 months.
6. Patients may not have received or plan to receive neoadjuvant systemic chemotherapy. 7) Patients unable to receive an aromatase inhibitor

8) Prior radiation to the affected breast 9) Previous cancers except for non-melanoma skin cancers or high risk cervical lesions in the past 5 years.

10) Previous breast cancer, tamoxifen, or aromatase inhibitor use. 11) Previous investigational immune therapy use-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women with resectable, non-metastatic breast cancer
Enrollment: 6 (Actual)
Dates: Start 2021-09-10 (Actual); Primary Completion 2023-06-16 (Actual); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants without the following safety events: TASAEs, persistent grade III/IV TAAEs, or toxicity-related delays in curative-intent surgery. Toxicity graded by CTCAE v5.0 and monitoring of AEs performed per FDA and NCI guidelines. | The safety assessment period begins with day 1 and ends within 30 days of surgical excision.
  yes/no outcome variable, ascertained for each individual subject, and reported as a binomial proportion for each arm. Safety will be reported for all subjects who receive at least one dose of drug/radiation/study therapy

SECONDARY OUTCOMES:
Immunogenicity of each therapeutic arm IFN-γ ELISPOT | throughout the study day 1, Day 8, Day 15, Day 29, Day 36, Week 7-9, Week 11, and 6 months post-surgery
  assessed by IFN-γ ELISPOT in PBMC
Immunogenicity of each therapeutic arm GEO-Mx digital spatial profiler | throughout the study day 1, Day 8, Day 15, Day 29, Day 36, Week 7-9, Week 11, and 6 months post-surgery
  assessed by GEO-Mx digital spatial profiler evaluation of Formalin-Fixed, parafin-embedded (FFPE) tumor and TCRβ evaluation for surviving-specific T cells in the tumor

CONTACTS AND LOCATIONS:
Overall Officials: Sasha Stanton, MD, Principal Investigator — Providence Health & Services
Locations (1):
- Providence Portland Medical Center, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Prat A, Saura C, Pascual T, Hernando C, Munoz M, Pare L, Gonzalez Farre B, Fernandez PL, Galvan P, Chic N, Gonzalez Farre X, Oliveira M, Gil-Gil M, Arumi M, Ferrer N, Montano A, Izarzugaza Y, Llombart-Cussac A, Bratos R, Gonzalez Santiago S, Martinez E, Hoyos S, Rojas B, Virizuela JA, Ortega V, Lopez R, Celiz P, Ciruelos E, Villagrasa P, Gavila J. Ribociclib plus letrozole versus chemotherapy for postmenopausal women with hormone receptor-positive, HER2-negative, luminal B breast cancer (CORALLEEN): an open-label, multicentre, randomised, phase 2 trial. Lancet Oncol. 2020 Jan;21(1):33-43. doi: 10.1016/S1470-2045(19)30786-7. Epub 2019 Dec 11. PMID 31838010
- [Background] von Minckwitz G, Untch M, Blohmer JU, Costa SD, Eidtmann H, Fasching PA, Gerber B, Eiermann W, Hilfrich J, Huober J, Jackisch C, Kaufmann M, Konecny GE, Denkert C, Nekljudova V, Mehta K, Loibl S. Definition and impact of pathologic complete response on prognosis after neoadjuvant chemotherapy in various intrinsic breast cancer subtypes. J Clin Oncol. 2012 May 20;30(15):1796-804. doi: 10.1200/JCO.2011.38.8595. Epub 2012 Apr 16. PMID 22508812
- [Background] Ellis MJ, Suman VJ, Hoog J, Lin L, Snider J, Prat A, Parker JS, Luo J, DeSchryver K, Allred DC, Esserman LJ, Unzeitig GW, Margenthaler J, Babiera GV, Marcom PK, Guenther JM, Watson MA, Leitch M, Hunt K, Olson JA. Randomized phase II neoadjuvant comparison between letrozole, anastrozole, and exemestane for postmenopausal women with estrogen receptor-rich stage 2 to 3 breast cancer: clinical and biomarker outcomes and predictive value of the baseline PAM50-based intrinsic subtype--ACOSOG Z1031. J Clin Oncol. 2011 Jun 10;29(17):2342-9. doi: 10.1200/JCO.2010.31.6950. Epub 2011 May 9. PMID 21555689
- [Background] Smith IE, Dowsett M, Ebbs SR, Dixon JM, Skene A, Blohmer JU, Ashley SE, Francis S, Boeddinghaus I, Walsh G; IMPACT Trialists Group. Neoadjuvant treatment of postmenopausal breast cancer with anastrozole, tamoxifen, or both in combination: the Immediate Preoperative Anastrozole, Tamoxifen, or Combined with Tamoxifen (IMPACT) multicenter double-blind randomized trial. J Clin Oncol. 2005 Aug 1;23(22):5108-16. doi: 10.1200/JCO.2005.04.005. Epub 2005 Jul 5. PMID 15998903
- [Background] Ellis MJ, Suman VJ, Hoog J, Goncalves R, Sanati S, Creighton CJ, DeSchryver K, Crouch E, Brink A, Watson M, Luo J, Tao Y, Barnes M, Dowsett M, Budd GT, Winer E, Silverman P, Esserman L, Carey L, Ma CX, Unzeitig G, Pluard T, Whitworth P, Babiera G, Guenther JM, Dayao Z, Ota D, Leitch M, Olson JA Jr, Allred DC, Hunt K. Ki67 Proliferation Index as a Tool for Chemotherapy Decisions During and After Neoadjuvant Aromatase Inhibitor Treatment of Breast Cancer: Results From the American College of Surgeons Oncology Group Z1031 Trial (Alliance). J Clin Oncol. 2017 Apr 1;35(10):1061-1069. doi: 10.1200/JCO.2016.69.4406. Epub 2017 Jan 3. PMID 28045625
- [Background] Karn T, Ruckhaberle E, Hanker L, Muller V, Schmidt M, Solbach C, Gatje R, Gehrmann M, Holtrich U, Kaufmann M, Rody A. Gene expression profiling of luminal B breast cancers reveals NHERF1 as a new marker of endocrine resistance. Breast Cancer Res Treat. 2011 Nov;130(2):409-20. doi: 10.1007/s10549-010-1333-x. Epub 2011 Jan 4. PMID 21203899
- [Background] Luen SJ, Salgado R, Fox S, Savas P, Eng-Wong J, Clark E, Kiermaier A, Swain SM, Baselga J, Michiels S, Loi S. Tumour-infiltrating lymphocytes in advanced HER2-positive breast cancer treated with pertuzumab or placebo in addition to trastuzumab and docetaxel: a retrospective analysis of the CLEOPATRA study. Lancet Oncol. 2017 Jan;18(1):52-62. doi: 10.1016/S1470-2045(16)30631-3. Epub 2016 Dec 7. PMID 27964843
- [Background] Loi S, Sirtaine N, Piette F, Salgado R, Viale G, Van Eenoo F, Rouas G, Francis P, Crown JP, Hitre E, de Azambuja E, Quinaux E, Di Leo A, Michiels S, Piccart MJ, Sotiriou C. Prognostic and predictive value of tumor-infiltrating lymphocytes in a phase III randomized adjuvant breast cancer trial in node-positive breast cancer comparing the addition of docetaxel to doxorubicin with doxorubicin-based chemotherapy: BIG 02-98. J Clin Oncol. 2013 Mar 1;31(7):860-7. doi: 10.1200/JCO.2011.41.0902. Epub 2013 Jan 22. PMID 23341518
- [Background] Denkert C, Loibl S, Noske A, Roller M, Muller BM, Komor M, Budczies J, Darb-Esfahani S, Kronenwett R, Hanusch C, von Torne C, Weichert W, Engels K, Solbach C, Schrader I, Dietel M, von Minckwitz G. Tumor-associated lymphocytes as an independent predictor of response to neoadjuvant chemotherapy in breast cancer. J Clin Oncol. 2010 Jan 1;28(1):105-13. doi: 10.1200/JCO.2009.23.7370. Epub 2009 Nov 16. PMID 19917869
- [Background] Denkert C, von Minckwitz G, Darb-Esfahani S, Lederer B, Heppner BI, Weber KE, Budczies J, Huober J, Klauschen F, Furlanetto J, Schmitt WD, Blohmer JU, Karn T, Pfitzner BM, Kummel S, Engels K, Schneeweiss A, Hartmann A, Noske A, Fasching PA, Jackisch C, van Mackelenbergh M, Sinn P, Schem C, Hanusch C, Untch M, Loibl S. Tumour-infiltrating lymphocytes and prognosis in different subtypes of breast cancer: a pooled analysis of 3771 patients treated with neoadjuvant therapy. Lancet Oncol. 2018 Jan;19(1):40-50. doi: 10.1016/S1470-2045(17)30904-X. Epub 2017 Dec 7. PMID 29233559
- [Background] Bates GJ, Fox SB, Han C, Leek RD, Garcia JF, Harris AL, Banham AH. Quantification of regulatory T cells enables the identification of high-risk breast cancer patients and those at risk of late relapse. J Clin Oncol. 2006 Dec 1;24(34):5373-80. doi: 10.1200/JCO.2006.05.9584. PMID 17135638
- [Background] Stanton SE, Adams S, Disis ML. Variation in the Incidence and Magnitude of Tumor-Infiltrating Lymphocytes in Breast Cancer Subtypes: A Systematic Review. JAMA Oncol. 2016 Oct 1;2(10):1354-1360. doi: 10.1001/jamaoncol.2016.1061. PMID 27355489
- [Background] Rodel F, Hoffmann J, Distel L, Herrmann M, Noisternig T, Papadopoulos T, Sauer R, Rodel C. Survivin as a radioresistance factor, and prognostic and therapeutic target for radiotherapy in rectal cancer. Cancer Res. 2005 Jun 1;65(11):4881-7. doi: 10.1158/0008-5472.CAN-04-3028. PMID 15930309
- [Background] Lutsiak ME, Semnani RT, De Pascalis R, Kashmiri SV, Schlom J, Sabzevari H. Inhibition of CD4(+)25+ T regulatory cell function implicated in enhanced immune response by low-dose cyclophosphamide. Blood. 2005 Apr 1;105(7):2862-8. doi: 10.1182/blood-2004-06-2410. Epub 2004 Dec 9. PMID 15591121
- [Background] Ge Y, Domschke C, Stoiber N, Schott S, Heil J, Rom J, Blumenstein M, Thum J, Sohn C, Schneeweiss A, Beckhove P, Schuetz F. Metronomic cyclophosphamide treatment in metastasized breast cancer patients: immunological effects and clinical outcome. Cancer Immunol Immunother. 2012 Mar;61(3):353-62. doi: 10.1007/s00262-011-1106-3. Epub 2011 Sep 14. PMID 21915801
- [Background] Karkada M, Weir GM, Quinton T, Sammatur L, MacDonald LD, Grant A, Liwski R, Juskevicius R, Sinnathamby G, Philip R, Mansour M. A novel breast/ovarian cancer peptide vaccine platform that promotes specific type-1 but not Treg/Tr1-type responses. J Immunother. 2010 Apr;33(3):250-61. doi: 10.1097/CJI.0b013e3181c1f1e9. PMID 20445345
- [Background] Benedict SH, Yenice KM, Followill D, Galvin JM, Hinson W, Kavanagh B, Keall P, Lovelock M, Meeks S, Papiez L, Purdie T, Sadagopan R, Schell MC, Salter B, Schlesinger DJ, Shiu AS, Solberg T, Song DY, Stieber V, Timmerman R, Tome WA, Verellen D, Wang L, Yin FF. Stereotactic body radiation therapy: the report of AAPM Task Group 101. Med Phys. 2010 Aug;37(8):4078-101. doi: 10.1118/1.3438081. PMID 20879569
- [Background] Hughes E, Scurr M, Campbell E, Jones E, Godkin A, Gallimore A. T-cell modulation by cyclophosphamide for tumour therapy. Immunology. 2018 May;154(1):62-68. doi: 10.1111/imm.12913. Epub 2018 Mar 9. PMID 29460448
- [Background] Scurr M, Pembroke T, Bloom A, Roberts D, Thomson A, Smart K, Bridgeman H, Adams R, Brewster A, Jones R, Gwynne S, Blount D, Harrop R, Hills R, Gallimore A, Godkin A. Low-Dose Cyclophosphamide Induces Antitumor T-Cell Responses, which Associate with Survival in Metastatic Colorectal Cancer. Clin Cancer Res. 2017 Nov 15;23(22):6771-6780. doi: 10.1158/1078-0432.CCR-17-0895. Epub 2017 Aug 29. PMID 28855352
- [Background] Butterfield LH, Ribas A, Dissette VB, Amarnani SN, Vu HT, Oseguera D, Wang HJ, Elashoff RM, McBride WH, Mukherji B, Cochran AJ, Glaspy JA, Economou JS. Determinant spreading associated with clinical response in dendritic cell-based immunotherapy for malignant melanoma. Clin Cancer Res. 2003 Mar;9(3):998-1008. PMID 12631598
- [Background] Disis ML, Wallace DR, Gooley TA, Dang Y, Slota M, Lu H, Coveler AL, Childs JS, Higgins DM, Fintak PA, dela Rosa C, Tietje K, Link J, Waisman J, Salazar LG. Concurrent trastuzumab and HER2/neu-specific vaccination in patients with metastatic breast cancer. J Clin Oncol. 2009 Oct 1;27(28):4685-92. doi: 10.1200/JCO.2008.20.6789. Epub 2009 Aug 31. PMID 19720923
- [Background] McArthur HL, Diab A, Page DB, Yuan J, Solomon SB, Sacchini V, Comstock C, Durack JC, Maybody M, Sung J, Ginsberg A, Wong P, Barlas A, Dong Z, Zhao C, Blum B, Patil S, Neville D, Comen EA, Morris EA, Kotin A, Brogi E, Wen YH, Morrow M, Lacouture ME, Sharma P, Allison JP, Hudis CA, Wolchok JD, Norton L. A Pilot Study of Preoperative Single-Dose Ipilimumab and/or Cryoablation in Women with Early-Stage Breast Cancer with Comprehensive Immune Profiling. Clin Cancer Res. 2016 Dec 1;22(23):5729-5737. doi: 10.1158/1078-0432.CCR-16-0190. Epub 2016 Aug 26. PMID 27566765